CLINICAL TRIAL: NCT04535934
Title: Novel Approaches for Quantitative Assessment of Adherence
Acronym: Tracer Pilot
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-0332; R01AI122298 (NIH)
Record Dates: First submitted 2020-02-14; First posted 2020-09-02 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for DNA will be obtained at the Visit 1 visit for those who consent to testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1 dose/week followed by 4 doses/week: Directly observed dosing regimen with 2 mg adenine 5+ (five stable-labeled nitrogens) as follows: 1 dose/week followed by 4 doses/week. The duration of each dosing regimen will be approximately 12 weeks. A washout period of approximately 12 weeks will separates the dosing regimens.
  Interventions: Other: Adenine 5+ (five stable-labeled nitrogens)
- 3 doses/week followed by 7 doses/week.: Directly observed dosing regimen with 2 mg adenine 5+ (five stable-labeled nitrogens) as follows: 3 doses/week followed by 7 doses/week. The duration of each dosing regimen will be approximately 12 weeks. A washout period of approximately 12 weeks will separates the dosing regimens.
  Interventions: Other: Adenine 5+ (five stable-labeled nitrogens)

INTERVENTIONS:
Other: Adenine 5+ (five stable-labeled nitrogens) — taggant coencapsulated with an excipient
  Other Names: taggant

SUMMARY:
Approximately 12 adults subjects will be enrolled. Participants will be randomized to one of two directly observed dosing regimens with 2mg adenine 5+ (five stable-labeled nitrogens) as follows: 1 dose/week followed by 4 doses/week OR 3 doses/week followed by 7 doses/week. Each dose regimen will have a duration of approximately 12 weeks and will be separated by a 12-week washout period for a total study duration of approximately 36 weeks.

Dried blood spots (DBS) and whole blood will be collect weekly. Urine will be collected less frequently, about every 2 weeks. The ratio of ATP 5+ to naturally occurring ATP 2+ is dried blood spots will be the primary outcome, as adenine is phosphorylated to ATP in red blood cells. Breakdown products will be measured in urine.

Investigators will allow flexibility in terms of which days are used for dosing for the 1, 3, and 4 dose(s)/week regimens. This is scientifically justified as investigators expect a 20-30 day half-life of ATP 5+ in DBS.

DETAILED DESCRIPTION:
Approximately twelve healthy adult volunteers with no contraindicated medical conditions or medications will be recruited from CU/Denver and the surrounding community.

Participants will be randomized to one of 2 sequences consisting of two directly observed dosing regimens with 2mg adenine 5+ per dose, 1 dose/week followed by 4 doses/week or 3 doses/week followed by 7 doses/week. Each dose regimen will have a duration of approximately 12 weeks and will be separated by an approximately 12-week washout period for a total study duration of approximately 36 weeks. The rationale for this study design is several fold. First, the lower doses are given initially to minimize the potential effects of carry-over in the second regimen. Second, 1 to 7 doses/week encompass a wide range of simulated adherence rates to assess the promise of this taggant, adenine 5+, as an adherence biomarker. Third, the 12 week duration is designed to achieve ~90% of steady-state given an estimated half-life of 20-30 days.

ELIGIBILITY:
Inclusion:

1. Ambulatory 18-40 year old adults.
2. Ability to comply with study procedures, including directly observed dosing visits and availability and use of video streaming technology.

Exclusion:

1. Inability to give informed consent
2. Pregnancy or plan to become pregnant in the next 12 months or unwillingness to use birth control
3. Current breastfeeding
4. Active psychiatric illness, social condition, or alcohol/drug abuse that, in the opinion of the investigators, would interfere with study requirements.
5. GFR estimate < 60 ml/min (MDRD equation).
6. Total bilirubin and/or hepatic transaminases (ALT and AST) ≥ 2.5x upper limit of normal
7. Absolute neutrophil count ≤ 1,500/mm3, platelets count ≤ 100,000/mm3, or hemoglobin ≤ 10 g/dL.
8. Symptomatic hemoglobinopathies or active hemolysis.
9. Any laboratory value or uncontrolled medical conditions that, in the opinion of the investigators, would interfere with the study conditions such as, heart disease and/or cancer.
10. Any investigational agents within 30 days of enrollment.
11. Plan to donate blood or plasma during study enrollment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult participants with no contraindicated medical conditions or medications.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Ratio of ATP 5+ to ATP 2+ in DBS | 9 months
  Ratio of ATP 5+ to ATP 2+ in DBS following directly observed therapy with 2mg of adenine 5+ at 1, 3, 4, and 7 doses/week
Dose-proportionality ATP 5+ to ATP 2+ in DBS | 9 months
  Dose-proportionality to relate ATP 5+ to ATP 2+ in DBS with adherence rate.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Anderson, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado- Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared